CLINICAL TRIAL: NCT03773016
Title: Using Computer Technology to Enable Arts and Crafts for People With Dementia in Care Homes
Brief Title: Touchscreen Technology and Art for People With Dementia in Care Homes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 18080
Record Dates: First submitted 2018-11-26; First posted 2018-12-12 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-12

CONDITIONS: Mild Dementia; Moderate Dementia
Keywords: care home; visual art; app; touchscreen technology; dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: The intervention activity will consist of the cross-over use of two different visual art apps in touchscreen tablets with people with mild to moderate dementia that lives in care homes. The study will take place in a nursing home in Nottinghamshire and will involve 12 residents of the care home with dementia and up to 12 staff members that are involved in participants' care. Study data collection will take 8 weeks; four weeks will involve the execution of the intervention and four weeks for additional measurements (collect consent, screening and end measures). Participants will be split into two groups of 6 participants; each group will use one app for two weeks and then change to the other app for another 2 weeks. Participants will be supported to use the app twice a week, with a maximum of 8 individual sessions over the four weeks. The data collection will consist of the observation of the activity and on the use of dementia-specific instruments and questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art apps - Group 1 (A-B) (Experimental): Cross-over use of two different visual art apps on touchscreen tablets (App A and App B)
  Interventions: Behavioral: Art apps
- Art apps - Group 2 (B-A) (Experimental): Cross-over use of two different visual art apps on touchscreen tablets (App B and App A)
  Interventions: Behavioral: Art apps

INTERVENTIONS:
Behavioral: Art apps — Participants will be split into two groups of 6 participants; each group will use one app for two weeks and then change to the other app for another 2 weeks. Participants will be supported to use the app twice a week, with a maximum of 8 individual sessions over the four weeks. The intervention will be delivered to the participants at a quiet room in the care home by two co-investigators, one will be the facilitator, and the other one will be the observer. The intervention is a 30-minutes of individual sessions, with 10 minutes of app use. The additional 20 minutes will include the setup of the equipment and preparation of the participant at the beginning of the session; and questions for the participants at the end.

SUMMARY:
The prevalence of dementia is rapidly growing worldwide, affecting 46.8 million people in 2015. The 2014 Alzheimer's Society report estimated that 311,730 people with dementia were living in care homes in the United Kingdom (UK). In care homes, people are more likely to be socially isolated and experience a lack of stimulation. It has been argued that access to meaningful activities is of high importance. One strategy that may engage older people in enjoyable leisure activities is the use of touchscreen technology. Previous research has indicated that people with dementia and care staff reported positive experiences when using touchscreen technology, showing improvements in quality of life, relationships and interpersonal interaction. A possible way to engage people with dementia with touchscreen technology could be through the use of the visual arts. Preliminary evidence shows the use of arts with this population to be beneficial in reducing behavioural symptoms, depression and isolation and make people with dementia more able to express feelings. The use of visual art activities in touchscreen technology is a promising idea, as positive results from interventions using these activities independently can be found in scientific literature. This intervention will consist of the use of two different visual art apps on touchscreen tablets with people with dementia living in care homes. Study data collection will take 8 weeks; four weeks will involve the execution of the intervention and four weeks for measurements. Participants will be supported to use the app twice-weekly, with a maximum of 8 individual sessions. So far, very little research on the benefits of visual art interventions on touchscreen devices has been made. Thus, there is a need to have more research on this topic. This study will add to research on this field, and its results could be valuable to care staff and people with dementia.

DETAILED DESCRIPTION:
SCIENTIFIC JUSTIFICATION:

People with dementia that live in care homes are more prone to experience a lack of stimulation and be socially isolated. Activities that are likely to be beneficial for people with dementia are social and leisure activities, as the activities promote engagement and improve affect. It has been argued that these activities should be of high importance in care settings and that care home residents living with dementia should have access to meaningful activities and are supported when engaging with the activities.

The use of touchscreen technology is one strategy that may possibly engage older people in enjoyable leisure activities. In past research, people with dementia and staff reported positive experiences with the use of technology in previous research that evaluate the impacts of touchscreen technology in care homes. This same research also showed supportive evidence for the positive contribution of the touchscreen technology for improvements in quality of life, relationships and interpersonal interactions. A literature review from 2017 on the use of touchscreen technology by people with dementia and its impact on wellbeing also shows supportive evidence for the use of touchscreen technology in dementia care. The researchers concluded that touchscreen-based interventions could provide benefits on mood, mental health, social interaction, quality of interaction, and sense of mastery. If people with dementia have the appropriate support for the use of touchscreen technology, it is evidently possible for people to benefit from its use.

A possible way to engage people with dementia with touchscreen technology could be through the use of the visual arts. Preliminary evidence shows that use of arts for people with dementia appears to be beneficial in reducing behavioural symptoms, depression and isolation and make people with dementia more able to express feelings. The use of visual art activities in touchscreen technology is a promising idea, as positive results from interventions using these activities separately can be found in scientific literature. So far, very little research on the benefits of visual art interventions on touchscreen devices has been made. Thus, there is a need to have more research on this topic. This study will add to research on this field and its results could be valuable to care staff and people with dementia. Providing people with dementia a set of exciting activities which have the potential to enrich people lives and be beneficial for wellbeing.

DESIGN AND METHODOLOGY:

The intervention activity will consist of the use of two different visual art apps on touchscreen tablets with people with mild to moderate dementia that lives in care homes. The study will take place in a nursing home in Nottinghamshire. It will involve 12 residents of the care home with dementia and staff members that are involved in participants' care. Potential participants will be identified by the care home staff, and staff members will indicate these people to the research team. Study data collection will take 8 weeks; four weeks will involve the execution of the intervention and four weeks for additional measurements (collect consent, screening and end measures). Given the nature of the intervention, no practical control condition would be a reasonable comparison for this intervention. Thus, the use of a cross-over design is a suitable control condition to be used in this study. Participants will be split into two groups of 6 participants; each group will use one app for two weeks and then change to the other app for another 2 weeks. Participants will be supported to use the app twice a week, with a maximum of 8 individual sessions over the four weeks. The data collection will consist of the observation of the activity and on the use of dementia-specific instruments and questionnaires.

This research aims to explore the supported use of two digital art apps in a participatory artistic activity with people living with dementia in residential care. The research team is interested in checking the efficacy of the activity. The team will also evaluate if art activities on touchscreen tablets are accepted by participants and carers and if the intervention is feasible in care settings.

The following research questions were formulated for this study:

What effects do participatory digital art on touchscreen tablets have on people with dementia in care homes? (impact on participants - efficacy)

How the insertion of the digital art activity is perceived by people with dementia and the care staff (acceptability of the intervention)

How can digital art apps be implemented in care homes to be delivered by the staff? (practicality of the intervention).

STUDY PROCESS AND TIMETABLE:

• Week 1 to Week 3:

These weeks will focus on:

Visits to explain the study to participants and consultees (30 minutes). Collection of the consent of the participants and consultees and answer questions (20 minutes).

Once the informed consent is signed potential participants with dementia will be accessed for cognition with the Montreal Cognitive Assessment - MoCA to ensure that the potential participants fit the inclusion criteria and will give the investigators a baseline on participants' cognition before the intervention (10 minutes).

Once the participants are selected, staff members will be contacted to reply to questions and questionnaires about the participant with dementia. Staff members will be asked to provide demographic information about the participants (3 minutes for each participant with dementia), to answer questions about the care home life (5 minutes), and to answer a proxy-instrument, the QUALIDEM for each of the participants (5 minutes for each participant with dementia).

Week 4 to Week 7:

The intervention activities with the participants with dementia will take place during these four weeks. The intervention will be delivered to the participants with dementia at a quiet room in the care home by two co-investigators, one will be the facilitator, and the other one will be the observer. All the sessions will be video recorded and analysed by two independent co-investigators. The use of video was preferred to observation and note taken as with it is possible to analyse the interaction between the participant and facilitator with the touchscreen tablet at the same time. With the analysis of the intervention through videos is also possible to focus on details that could be missed with observations, as videos give the opportunity to pause and repeat key points of the interaction for a comprehensive analysis.

The intervention is a 30-minutes of individual sessions, with 10 minutes of app use. The additional 20 minutes will include the setup of the equipment and preparation of the participant at the beginning of the session; and questions for the participants at the end. The sessions will happen in the afternoon four days a week (on weekdays), with 6 participants per day (one of the groups). Each group will have fixed session days, to make the staff aware of which participants would have a session on a specific day.

Data collection here will be made through:

Participants' observation: Participants' behaviour in the video records of the sessions will be analysed with an adapted version of the Greater Cincinnati Chapter Wellbeing Observation Tool.

Questions to participants: At the end of each session, the participants will be asked to answer questions on visual analogue scales (VAS) to evaluate participants subjective wellbeing at that moment (3 minutes).

Questionnaires and questions to staff: Staff members will be asked to answer the QUALIDEM once a week during the 4-week intervention for each of the participants (5 minutes for each participant with dementia).

The research team will also evaluate the acceptability and practicality of the intervention:

Acceptability: Participants will be asked at the end of the sessions (once a week) questions about satisfaction with the apps and the intervention (3 minutes) relevance of the activity, and if would be interest in continue the use of the apps (VAS, and open questions). The research team will also check for actual use of the touchscreen tablet between the sessions and will provide a form to the care staff keep a record (1 minute for each entry).

Practicality: To evaluate the practicality of the intervention, the participants and the staff will be asked on the opinion on frequency and duration of the intervention (ideal and what was received) (3 minutes). During the intervention the researchers will make observations on care home daily life and will collect information on the type and amount of resources needed, training required and time to support the intervention. There also will be an analysis of the barriers and facilitators for the implementation of the activity in care homes. One of the researchers will collect this information through field notes of observation of the sessions and discussions with the care staff.

Week 8:

For end measurements, the MoCA (10 minutes) will be used with participants with dementia and the staff members will be asked to answer the QUALIDEM for each of the participants (5 minutes for each participant with dementia).

• At a later point (data collection finished): Once data collection is complete, the research team will develop the guidance on the use of touchscreen tablets in residential care for people with dementia. Staff members from the care home will be asked to give feedback on the guidance through informal consultation. This informal consultation could happen through email communication or in-person meetings. This should happen within 2 months after the end of data collection. The analysis and writing up findings should take up to 5 months.

ELIGIBILITY:
Inclusion Criteria:

Participants with dementia:

* To be living in a Care Home in Nottinghamshire;
* To have mild dementia [21 to 26 points in the Mini-Mental State Examination (MMSE) or a comparable score on the MoCA from 16 to 20 points] or moderate dementia [10 to 20 points on the MMSE or a comparable score on the MoCA from 2 to 15 points];
* To be willing to use apps on touchscreen tablets;
* Ability to give informed consent or have a consultee that provides advice;
* Ability to speak and understand English.

Nursing home staff:

* To be involved in the care of at least one of the participants;
* Ability to speak and understand English.

Exclusion Criteria:

Participants with dementia:

* To have conditions that could limit hand-control (e.g. stroke, Parkinson's disease);
* To have severe visual or hearing impairments;
* Simultaneous participation in any other interventional study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-04-12 (Estimated); Study Completion 2019-04-12 (Estimated)

PRIMARY OUTCOMES:
Change on Wellbeing | 1 month
  Assessed by Greater Cincinnati Chapter Wellbeing Observation Tool (observational tool to evaluate wellbeing during art interventions) - 19 items with domains of wellbeing and ill-being. Each item can be scored from 0 (never) to 4 (always).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Astell AJ, Joddrell P, Groenewoud H, de Lange J, Goumans M, Cordia A, Schikhof Y. Does familiarity affect the enjoyment of touchscreen games for people with dementia? Int J Med Inform. 2016 Jul;91:e1-8. doi: 10.1016/j.ijmedinf.2016.02.001. Epub 2016 Feb 12. PMID 26897552
- [Background] Brooker DJ, Woolley RJ, Lee D. Enriching opportunities for people living with dementia in nursing homes: an evaluation of a multi-level activity-based model of care. Aging Ment Health. 2007 Jul;11(4):361-70. doi: 10.1080/13607860600963679. PMID 17612800
- [Background] Cohen-Mansfield J, Dakheel-Ali M, Thein K, Marx MS. The impact of stimulus attributes on engagement of nursing home residents with dementia. Arch Gerontol Geriatr. 2009 Jul-Aug;49(1):1-6. doi: 10.1016/j.archger.2008.04.002. Epub 2008 Jul 7. PMID 18602707
- [Background] Dichter, M., Ettema, T., Schwab, C., Meyer, G., Bartholomeyczik, S., Halek, M., & Dröes, R. (2016). QUALIDEM-user guide. DZNE/VUmc, Witten/Amsterdam.
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Gross SM, Danilova D, Vandehey MA, Diekhoff GM. Creativity and dementia: does artistic activity affect well-being beyond the art class? Dementia (London). 2015 Jan;14(1):27-46. doi: 10.1177/1471301213488899. Epub 2013 May 22. PMID 24339088
- [Background] Han, A., Radel, J., McDowd, J. M., & Sabata, D. (2016). The Benefits of Individualized Leisure and Social Activity Interventions for People with Dementia: A Systematic Review. Activities, Adaptation & Aging, 40(3), 219-265. doi:10.1080/01924788.2016.1199516
- [Background] Hannemann BT. Creativity with dementia patients. Can creativity and art stimulate dementia patients positively? Gerontology. 2006;52(1):59-65. doi: 10.1159/000089827. PMID 16439826
- [Background] Joddrell, P. (2017). Investigating the potential of touchscreen technology to create opportunities for independent activity with people living with dementia. University of Sheffield.
- [Background] Joddrell, P., Hernandez, A., & Astell, A. J. (2016). Identifying Existing, Accessible Touchscreen Games for People Living with Dementia. Computers Helping People with Special Needs, Icchp 2016, Pt I, 9758, 509-514. doi:10.1007/978-3-319-41264-1_69
- [Background] Kinney JM, Rentz CA. Observed well-being among individuals with dementia: Memories in the Making, an art program, versus other structured activity. Am J Alzheimers Dis Other Demen. 2005 Jul-Aug;20(4):220-7. doi: 10.1177/153331750502000406. PMID 16136845
- [Background] Leng FY, Yeo D, George S, Barr C. Comparison of iPad applications with traditional activities using person-centred care approach: impact on well-being for persons with dementia. Dementia (London). 2014 Mar 1;13(2):265-73. doi: 10.1177/1471301213494514. Epub 2013 Jul 19. PMID 24339097
- [Background] Leuty V, Boger J, Young L, Hoey J, Mihailidis A. Engaging older adults with dementia in creative occupations using artificially intelligent assistive technology. Assist Technol. 2013 Summer;25(2):72-9. doi: 10.1080/10400435.2012.715113. PMID 23923689
- [Background] Mihailidis, A., Blunsden, S., Boger, J., Richards, B., Zutis, K., Young, L., & Hoey, J. (2010). Towards the development of a technology for art therapy and dementia: Definition of needs and design constraints. The Arts in Psychotherapy, 37(4), 293-300.
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] NICE. (2011). Donepezil, galantamine, rivastigmine and memantine for the treatment of Alzheimer's disease. Retrieved from https://www.nice.org.uk/guidance/ta217
- [Background] Smith, S. K. (2015). Exploring the potential of touch-screen computer technology in promoting enjoyable activities with people living with dementia: A visual ethnography. University of Sheffield.
- [Background] Trzepacz PT, Hochstetler H, Wang S, Walker B, Saykin AJ; Alzheimer's Disease Neuroimaging Initiative. Relationship between the Montreal Cognitive Assessment and Mini-mental State Examination for assessment of mild cognitive impairment in older adults. BMC Geriatr. 2015 Sep 7;15:107. doi: 10.1186/s12877-015-0103-3. PMID 26346644
- [Background] Tyack C, Camic PM. Touchscreen interventions and the well-being of people with dementia and caregivers: a systematic review. Int Psychogeriatr. 2017 Aug;29(8):1261-1280. doi: 10.1017/S1041610217000667. Epub 2017 Apr 27. PMID 28446258
- [Background] Tyack C, Camic PM, Heron MJ, Hulbert S. Viewing Art on a Tablet Computer: A Well-Being Intervention for People With Dementia and Their Caregivers. J Appl Gerontol. 2017 Jul;36(7):864-894. doi: 10.1177/0733464815617287. Epub 2015 Dec 16. PMID 26675353
- [Background] Upton, D., Upton, P., Jones, T., Jutlla, K., Brooker, D., & Grove, H. (2011). Evaluation of the impact of touch screen technology on people with dementia and their carers within care home settings. UK: University of Worcester.